CLINICAL TRIAL: NCT02511847
Title: An Open Label, Phase II Trial of Afatinib With Paclitaxel for the Neoadjuvant Treatment of Triple-Negative Breast Cancer and Research of Biomarkers of Activity and Efficacy of Afatinib
Brief Title: Trial of Afatinib With Paclitaxel for Neoadjuvant Therapy of TNBC and Research of Biomarkers of Afatinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201408024MIPC
Record Dates: First submitted 2015-07-16; First posted 2015-07-30 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast Cancer; EGFR; Afatinib; Paclitaxel; Pathologic complete remission
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Pathologic Complete Response | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm (Other): Drug: Afatinib (single group assignment)
  1. First phase: Afatinib montherapy
  2. The following phases: combination with oral afatinib and weekly paclitaxel in a 3-weekly course for total of four courses.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 1. Afatinib 40 mg per day for 14 days, then evaluation, every subject will go into the following phase no matter whether she had response or not
  2. Afatinib 40 mg per day, day 1 to day 21, in combination with paclitaxel 80 mg/m² on days 1, 8, 15 in a 3-weekly course.

SUMMARY:
[Background]: Triple-negative breast cancer (TNBC) is defined by a lack of expression of both estrogen and progesterone receptor as well as human epidermal growth factor receptor 2 (HER-2). TNBC is characterized by distinct molecular, histological and unfavorable clinical features despite the high rates of response to chemotherapy. Based on the above reasons, it is important to emergently develop novel therapies and/or treatment strategies to increase treatment efficacies and the survival rate of TNBC.

[Rationale]: Overexpression of epidermal growth factor receptor (EGFR/ErbB1) and EGFR mutation have been reported in TNBC and may therefore be a valid target for anti-tumor therapy in TNBC. Afatinib (BIBW 2992) is an ErbB-family blocker that irreversibly inhibits signaling from all relevant ErbB-family dimers. Afatinib has demonstrated preclinical activity in triple-negative breast cancer cell lines and xenograft models of breast cancer, and clinical activity in phase I studies. Based on the assumption that uncontrolled ErbB-signaling is directly related to an increased oncogenic potential in TNBC, the studying afatinib in the neoadjuvant treatment of TNBC patients is important and provides a novel therapy.

[Aims] The primary endpoint is to evaluate the pathologic complete response of the combination of afatinib and weekly paclitaxel in TNBC patients receiving neoadjuvant treatment. The secondary endpoints are to evaluate the clinical response and safety of afatinib with and without paclitaxel, and to explore the different afatinib-affecting downstream molecular pathways as well as potential biomarkers predicting the response of afatinib with and without paclitaxel.

[Patients and methods]: Patients with TNBC (clinical T2-T3, N0-N1, M0; clinical T1-3, N1-2, M0; or any T4a tumor) and received neoadjuvant treatment will included in this open, label, multi-center phase II study. Our schema is as follows: (1) Afatinib 40 mg per day for 14 days, then evaluation, every subject will go into the following phase no matter whether she had response or not (2) the following phase (the combination with afatinib and paclitaxel): Afatinib 40 mg per day, day 1 to day 21, in combination with paclitaxel 80 mg/m² on days 1, 8, 15 in a 3-weekly course. In addition to the clinical assessment, we will evaluate the potential predictive biological markers of activity of Afatinib with and without paclitaxel and dynamic changes of molecular makers ([serum and tissue samples: before treatment, 2 weeks after treatment, and operation timing]; potential molecules, such as EGFR, EGFR-signaling, FGFR, FGFR-signaling, ERK, p53, NF-κB, and etc. were evaluated through the immunohistochemical stains, mutation analysis, mRNA [RT-PCR], single nucleotide polymorphism analysis, and FISH analysis). In addition, the genetic expression profiles will be compared between afatinib-responsive and afatinib-unresponsive samples.

[Expected Results]: The promising clinical activity, tolerable toxicity, and potential biomarkers of afatinib with and without paclitaxel in TNBC patients receiving neoadjuvant setting will be demonstrated. The results from this study can be used to conduct a larger trial that would allow us to confirm or validate the hypotheses generated.

DETAILED DESCRIPTION:
Objects: Phase II study

Primary Objective :

To evaluate the efficacy of combination of afatinib and weekly paclitaxel as assessed by pathologicalresponse in the residual tumor.

Secondary Objectives:

1. Efficacy of afatinib as assessed by the ultrasound of the breast.
2. Adverse effect of afatinib monotherapy and the combination of afatinib and weekly paclitaxel.
3. Correlation between baseline potential biomarkers and radiological response of afatinib monotherapy.
4. Correlation between down- or up-regulation of potential biomarkers (in pre-treatment biopsy and surgical specimen) and radiological response to afatinib and paclitaxel.
5. To identify the pharmacodynamic biomarkers, the following translational researches will be carried out on initial tumor biopsy and surgical specimen.
6. To evaluate the dynamic changes of circulating tumor cells and cell-free DNA after afatinib monotherapy and after the combination of afatinib and weekly paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age ≥20 years
2. Histologically confirmed invasive ER-, PR-, and HER2-negative (triple-negative) adenocarcinoma of the breast
3. Triple-negative tumors are defined as:

   i. For HER2-negative: Fluorescence in situ hybridization (FISH)-negative (defined by ratio <2.0) or Immunohistochemical (IHC) 0, IHC 1+, or IHC 2+ or IHC 3+and FISH-negative (defined by ratio <2.0) ii. For ER- and PR-negative: < 5% tumor staining by immunohistochemistry (IHC)
4. The first TNBC 20 patients with or without EGFR expression or mutation are eligible. Interim analysis of response rate will be calculated to determine the criteria of 21 to 40 patients.
5. All of the newly diagnosed TNBC patients should be met the following criteria: clinical node-positive with any T stage patents or clinical node-negative patients with cT2-4. cT1N0M0 lesions are excluded. Patients with metastatic disease are excluded. The measurement method of tumor size can be by physical exam and/or image study.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
7. Within 2 weeks prior randomization:

   i. Adequate bone marrow function, hepatic function, and renal function. ii. Controlled blood pressure with or without antihypertensive treatment iii. Normal prothrombin time (PT) and partial thromboplastin time (PTT) iv. Adequate cardiac function assessed by 12-lead ECG and if clinically indicated echocardiography to document LVEF
8. Bilateral, synchronous breast cancer is allowed if one primary tumor meets the inclusion criteria.
9. Adequate bone marrow function defined as WBC ≥3.5 x 109/L, ANC ≥1.5 x 109/L, platelets ≥LLN, and hemoglobin ≥10 g/dL.
10. Adequate liver function defined as total serum bilirubin ≤1.5X ULN and serum transaminases ≤2.5X ULN
11. Adequate renal function defined as creatinine ≤1.5X ULN
12. Able and willing to give informed consent and comply with the protocol
13. Written informed consent obtained prior to any Screening/baseline procedures
14. Knowledge of the investigational nature of the study and ability to provide consent for study participation; and ability and willingness to comply with study visits, treatment, testing, and other study procedures

Exclusion Criteria:

1. ER+ (>5%) or PR+ (>5%) or Her-2 overexpression
2. Active second malignancy during the last five years except non melanomatous skin cancer or carcinoma in situ of the cervix.
3. Prior chemotherapy, radiotherapy or targeted therapy including afatinib or Her-2 or EGFR inhibitors.
4. Participation in another interventional clinical trial in the preceding 30 days prior to trial.
5. Patients with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study
6. Prior hypersensitivity reactions to a taxane or to Cremophor® EL (polyoxyethylated castor oil)
7. Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive β-HCG laboratory test (serum > 5 mIU/mL)
8. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 180 days after study treatment. Highly effective contraception methods include:

   * True abstinence in line with the preferred and usual lifestyle of the subject
   * Female subject or male partner sterilization or
   * Combination of any two of the following (a+b or a+c, or b+c):

     1. Use of oral, injected or implanted hormonal methods of contraception
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
     3. Barrier methods of contraception: condom for male partner or occlusive cap
     4. (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
9. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of pathologic response of the combination of afatinib and weekly paclitaxel | 2 years
  Evaluation of the pathologic complete response of the combination of afatinib and weekly paclitaxel in TNBC patients with neoadjuvant treatment.

SECONDARY OUTCOMES:
Efficacy of afatinib | 2 years
  The radiologic response will be assessed on ultrasound of the breast.
Adverse effect of afatinib monotherapy and the combination of afatinib and weekly paclitaxel | 2 years
Correlation between potential biomarkers and radiological response of afatinib montherapy | 2 years
Correlation between down- or up-regulation of potential biomarkers and radiological response to afatinib and paclitaxel | 2 years
Identification of the pharmacodynamic biomarkers by initial tumor biopsy and surgical specimen | 2 years
Evaluation of the dynamic changes of circulating tumor cells and cell-free DNA after afatinib monotherapy and after the combination of afatinib and weekly paclitaxel | 2 years
  circulating tumor cells is a new technigue compatible with cell search.

CONTACTS AND LOCATIONS:
Overall Officials: Chiun-Sheng Huang, PhD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan